CLINICAL TRIAL: NCT04172272
Title: The Influence of the Transversus Abdominis Plane Block on the Intensity of Postoperative Pain and the Concentration of Proinflammatory and Pain Factors After Laparotomy for Gynecological Procedures
Brief Title: The Influence of TAP Block in the Control of Postoperative Pain After Laparotomy for Gynecological Procedures
Acronym: TAP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: General Hospital Pula (Other)
Collaborators: Clinical Hospital Center Rijeka (Other)
Responsible Party: Principal Investigator, Tomislav Perkov, MD, Principal Investigator, General Hospital Pula
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 3
Record Dates: First submitted 2019-11-08; First posted 2019-11-21 (Actual); Last update posted 2019-11-21 (Actual); Status verified 2019-11

CONDITIONS: Leiomyoma; Pelvic Organ Prolapse; Abnormal Uterine Bleeding; Chronic Pain; Premalignant Lesion; Endometriosis
Keywords: Transversus abdominis plane block; Laparotomy; Hysterectomy; Postoperative pain; Cytokines; Visual analogue scale; Quality of recovery
MeSH Terms: conditions — Leiomyoma; Pelvic Organ Prolapse; Metrorrhagia; Chronic Pain; Endometriosis; Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Systemic multimodal analgesia only (Active Comparator): In the first group, patients will receive intravenous, systemic, multimodal analgesia: paracetamol 1 gram and ketoprofen 100 mg every 8 hours for 24 hours. Analgesia will start immediately after surgery. If the pain persists, the patient will be given "rescue" analgesia: tramadol 50 mg intravenously up to a maximum dose of 400 mg / 24 h and other analgesics if needed.
  Interventions: Drug: Systemic multimodal analgesia administered intravenously
- TAP block only (Experimental): In the second group there will be patients in who will be given the TAP block. The TAP block will be given postoperatively before waking. It will be given bilaterally in the before mentioned anatomic region (the so-called lateral TAP block) of 0.25% levobupivacaine in 40 ml bilaterally. If such analgesia is not satisfactory, tramadol 50 mg intravenously, up to a maximum dose of 400 mg / 24h, and other analgesics will be given at the request of the patient.
  Interventions: Procedure: Transversus abdominis plane block (TAP block)
- Combined TAP block with systemic multimodal analgesia (Experimental): In the third group there will be patients who will be treated with TAP block in addition to systemic, mutimodal analgesia. If such analgesia is not satisfactory, tramadol 50 mg intravenously, up to a maximum dose of 400 mg / 24h, and other analgesics will be given at the request of the patient.
  Interventions: Other: Combined transversus abdominis plane block (TAP block) with systemic multimodal analgesia administered intravenously

INTERVENTIONS:
Drug: Systemic multimodal analgesia administered intravenously — Paracetamol 1 gram and ketoprofen 100 mg every 8 hours for 24 hours. Analgesia will start immediately after surgery. If the pain persists, the patient will be given "rescue" analgesia: tramadol 50 mg intravenously up to a maximum dose of 400 mg / 24 h and other analgesics if needed.
  Arms: Systemic multimodal analgesia only
Procedure: Transversus abdominis plane block (TAP block) — The TAP block will be given postoperatively before waking. It will be given bilaterally in the before mentioned anatomic region (the so-called lateral TAP block) of 0.25% levobupivacin in 40 ml bilaterally. If the pain persists, the patient will be given "rescue" analgesia: tramadol 50 mg intravenously up to a maximum dose of 400 mg / 24 h and other analgesics if needed.
  Arms: TAP block only
Other: Combined transversus abdominis plane block (TAP block) with systemic multimodal analgesia administered intravenously — TAP block in addition to systemic, mutimodal analgesia. If such analgesia is not satisfactory, tramadol 50 mg intravenously, up to a maximum dose of 400 mg / 24h, and other analgesics will be given at the request of the patient.
  Arms: Combined TAP block with systemic multimodal analgesia

SUMMARY:
This study evaluates the influence of the transversus abdominis plane block on the intensity of postoperative pain and the concentration of proinflammatory and pain factors after hysterectomy by laparotomy. The patients will be randomized in three groups.In the first group, patients will receive intravenous, systemic, multimodal analgesia.In the second group there will be patients in who will be given the TAP block. The TAP block will be given postoperatively before waking. It will be given bilaterally in the before mentioned anatomic region (the so-called lateral TAP block). In the third group there will be patients who will be treated with TAP block in addition to systemic, mutimodal analgesia. The research will be based on completing a questionnaire (VAS scale and QoR questionnaire) and taking peripheral blood out. We expect that the concentration of proinflammatory and pain factors in patients treated with a TAP block will be lower and the quality of recovery will be better than that of patients receiving standard analgesic therapy (systemic multimodal analgesia).

DETAILED DESCRIPTION:
The influence of the transversus abdominis plane block on the intensity of postoperative pain and the concentration of proinflammatory and pain factors after laparotomy for gynecological procedures

Showing the problem

Hysterectomy is one of the most commonly performed surgical operations. Indications for hysterectomy are numerous and include benign and malignant etiology. Symptomatic leiomyomas, pelvic organ prolapse, abnormal uterine bleeding, endometriosis, chronic pain, and premalignant lesions are the most commonly benign indications for hysterectomy. The uterus can be removed using an abdominal, vaginal or laparoscopic approach. Each of these approaches is related to postoperative pain as well as on an increase in inflammatory factors that may adversely affect the recovery of patients. Therefore, pain management has become one of the major quality of life issues in the postoperative period. Post-operative pain is not only a limitation for the patient but the long-term pain can have deleterious effects on respiratory, cardiocirculatory and neuroendocrine function. Adverse physiological changes due to inadequate or insufficient postoperative analgesia can lead to increased morbidity and mortality to the patients.

The main assumption of the so-called "preventive analgesia" is to try to prevent the influx of nociceptive stimuli (surgical trauma) to the spinal cord and thus reduce postoperative pain. For this purpose, various anesthesiologic regional techniques (epidural analgesia, transversus abdominis plane block) are used for trying to reduce the activation of postoperative pain. Timely application of "preventive analgesia" and its long enough and intense action are essential as they could be captured all afferent nociceptive impulses. In the choice of optimal analgesia, the type and location of the procedure, the duration of the analgesic therapy required, individual risk factors and contraindications are of great importance. Preventive analgesia may be initiated immediately before the onset of tissue injury (eg epidural or spinal analgesia), immediately after surgery using regional blocks or intravenous analgesia for a well-defined period of time (eg at intervals of 3 to 6 hours). The goal of quality treatment of acute pain is not only optimal analgesia, but also for reducing complications. One of the newer techniques for postoperative analgesia is a transversus abdominis plane block (TAP), which is part of regional anesthesia techniques. It is a peripheral nerve block that blocks nerves located in the fascia layer between the m. transversus abdominis and the m. obliqus internus, which innervate the anterolateral abdominal wall. These nerves include the intercostal (Th7-Th11), subcostal (Th12), iliohypogastric and ilioinguinal (L1) nerves. A local anesthetic administered in the layer between the m. transversus abdominis and the m. obliqus internus results in anesthesia of the anterolateral abdominal wall. This technique achieves analgesia of the skin, subcutaneous, muscle, and parietal peritoneum in a given region. The blockage of these nerves is useful primarily for postoperative analgesia after abdominal surgery, including gynecologal too.

In major surgical procedures such as uterine removal (hysterectomy), pain and stress caused by surgical tissue injury stimulate a strong pro-inflammatory response, so establishing effective postoperative analgesia which adequately relieved the pain is of great importance. In this study, investigators will evaluate the effect of a transversus abdominis plane block on the severity of postoperative pain as well as its effect on proinflammatory and pain factors in patients following gynecologic surgery performed with a laparotomy approach. The investigators will also compare the use of standard systemic multimodal analgesia and the TAP block (as well as their combination) in the control of postoperative pain. Studies have shown that both approaches are effective in controlling postoperative pain, but comparative studies are rare, and none has so far examined the concentration of proinflammatory and pain factors in operated patients.

Hypothesis

The basic hypothesis is that a transversus abdominis plane block reduces postoperative pain in patients after gynecologic surgery performed with a laparotomic approach. The expectation is that the concentration of proinflammatory and pain factors in patients treated with a TAP block will be lower and the quality of recovery will be better than that of patients receiving standard analgesic therapy (systemic multimodal analgesia).

Objectives of the research

1. Compare the three forms of postoperative analgesia dividing patients in the three groups (TAP block only, systemic multimodal analgesia only and combined TAP block with systemic multimodal analgesia) after gynecological surgeries to show which one has the highest value in controlling postoperative pain.
2. Analyze the impact of the TAP block on postoperative pain, using a visual analogue scale (VAS) in patients after gynecological surgery.
3. Analyze the impact of TAP block combined with systemic, multimodal analgesia on postoperative pain, using the VAS scale, in patients after gynecological surgery.
4. Analyze the concentration of proinflammatory cytokines and pain factors (IL-1ß, IL-6, cortisol, catecholamines) in the plasma of patients who will receive a TAP block after gynecological surgery.
5. Analyze the impact of the TAP block on the quality of recovery, measured with quality of recovery (QoR) questionnaire in patients after gynecological surgery.
6. Correlate values of subjective assessment of postoperative pain intensity using VAS scale with concentration of proinflammatory and biomarkers for pain (IL-1ß, IL-6, cortisol, catecholamines) in patients in whom postoperative pain after gynecological surgery will be treated with TAP block or systemic multimodal analgesia.

Construction of the study

The structure will be a prospective, randomized, single-blind study.

Subjects (Material)

The number of women enrolled in the study will be 75. Patients will be interviewed in detail prior to surgery to be informed of planned anesthesia, surgery and postoperative pain control, and will sign informed consent and consent to participate in the study.

From each patient by standard technique venous blood will be taken out from peripheral vein at certain intervals after surgery. The patients will be asked by the examiner to complete VAS scale or and the QoR questionnaire.

Methods

Hysterectomy and / or adnexectomy will be performed in patients included in the study due to benign gynecological pathology with a laparotomy approach. Baseline patient data will be determined based on a detailed medical history and medical records, clinical examination of each patient and imaging tests. A definitive diagnosis of benign gynecological pathology will be obtained after a histopathological analysis of the tissue. A detailed interview will be done with the patients before surgery, and patients will be informed about the planned anesthesia, surgery and postoperative pain control. After that patients will sign an informed consent and the consent for participating in the study. For the purpose of the study, patients will be randomized into three groups regarding to the treatment technique for postoperative pain. The doctor ( researcher) will, by the computer program Datlnf Ranolist do the randomization. So that way the researcher will determine the type of analgesia the patient will receive. In the first group, patients will receive intravenous, systemic, multimodal analgesia: paracetamol 1 gram and ketoprofen 100 mg every 8 hours for 24 hours. Analgesia will start immediately after surgery. If the pain persists, the patient will be given "rescue" analgesia: tramadol 50 mg intravenously up to a maximum dose of 400 mg / 24 h and other analgesics if needed. In the second group there will be patients in who will be given the TAP block. The TAP block will be given postoperatively before waking. It will be given bilaterally in the before mentioned anatomic region (the so-called lateral TAP block) of 0.25% levobupivacin in 40 ml bilaterally. If such analgesia is not satisfactory, tramadol 50 mg intravenously, up to a maximum dose of 400 mg / 24h, and other analgesics will be given at the request of the patient. In the third group there will be patients who will be treated with TAP block in addition to systemic, mutimodal analgesia. If such analgesia is not satisfactory, tramadol 50 mg intravenously, up to a maximum dose of 400 mg / 24h, and other analgesics will be given at the request of the patient. The standardized protocol will determine the general information of each patient to be included in the study: ID, age and gender. 25 patients will be included in each group. The research will be based on completing a questionnaire (VAS scale and QoR questionnaire) and taking peripheral blood out. Blood will be taken from the peripheral vein by standard technique in a volume of 10 ml before surgery and 6, 24 and 48 hours after surgery. VAS scale (at rest and in motion) will be determined before surgery and 3, 6, 12, 24 and 48 hours after surgery. The QoR questionnaire will be examined before surgery, 24 hours after surgery and 30 days after surgery. The concentrations of individual cytokines (IL-1ß, IL-6) and hormones (catecholamines, cortisol) related to inflammation and pain will be determined by standard laboratory methods from peripheral blood. Cytokine and hormone concentrations will be determined by enzyme immunofluorescence method according to the manufacturer's instructions. All results obtained through the questionnaire or blood test will only serve for the purpose of the study and will not have diagnostic, therapeutic or prognostic value for the patients included in the study.

Statistical methods

Statistical data processing will be performed in the Statistica 12.0 computer program (StatSoft, Inc., Tulsa, OK, USA). When calculating differences between experimental groups, investigators will use the Kruskal Walis ANOVA nonparametric test for small independent samples. Changes will be considered statistically significant with p <0.05. We will use the Mann-Whitney U test subsequently to determine between which two of the more comparable groups there is statistical significance. Correlations will be examined by Pearson or Spearman correlation test, depending on the results of the data distribution analysis. Differences between variables expressed at nominal level will be examined using the chi-square test. Image and spreadsheet views of the results will be made in Microsoft Excel and Statistica 12.0.

Expected scientific contribution

It is hoped that the results of the proposed study will shed light on the impact of various anesthesiologic techniques (transversus abdominis plane block, intravenous systemic multimodal analgesia and their combination) on postoperative pain and the concentration of proinflammatory and pain factors after gynecologic surgery performed with a laparotomy approach. Investigators expect that the use of regional analgesia technique (TAP block) will lead to a reduction in postoperative pain and proinflammatory factors and pain factors examined, thereby contributing to a faster recovery and better outcome of their treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a benign gynecological condition, who underwent hysterectomy by laparotomy approach.

Exclusion Criteria:

* under aged
* pregnant women,
* patients with malignant gynecological disease,
* those with anesthesiologic risk of ASA III or more,
* persons who are hypersensitive to anesthetics and analgesics,
* patients who do not agree with the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 75 (Estimated)
Dates: Start 2019-09-24 (Actual); Primary Completion 2020-09-24 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
The impact of three forms of postoperative analgesia (TAP block, systemic multimodal analgesia, combined TAP block and systemic multimodal analgesia)on postoperative pain after gynecological surgery | 48 hours
  Self-reported pain intensity using a standard visual analogue scale (VAS, from 0 to 10) in patients after gynecological surgery.
Concentration of proinflammatory and pain factors in patients on postoperative pain after gynecological surgery | Before surgery and 6, 24 and 48 hours after surgery
  Change in concentrations of individual cytokines (IL-1ß, IL-6) and hormones (catecholamines, cortisol) related to inflammation and pain
Quality of recovery after gynecological surgery | 30 days
  The impact of three forms of postoperative analgesia (TAP block, systemic multimodal analgesia and combined TAP block and systemic multimodal analgesia) on the quality of recovery in patients after gynecological surgery, measured by using a widely accepted 40-item Quality of Recovery (QoR) questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Tomislav Perkov, MD, Principal Investigator — GH Pula
Locations (2):
- Croatia (2):
  - GH Pula, Pula
  - Clinical centre Rijeka, Rijeka

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Young MJ, Gorlin AW, Modest VE, Quraishi SA. Clinical implications of the transversus abdominis plane block in adults. Anesthesiol Res Pract. 2012;2012:731645. doi: 10.1155/2012/731645. Epub 2012 Jan 19. PMID 22312327
- [Background] McDonnell JG, O'Donnell B, Curley G, Heffernan A, Power C, Laffey JG. The analgesic efficacy of transversus abdominis plane block after abdominal surgery: a prospective randomized controlled trial. Anesth Analg. 2007 Jan;104(1):193-7. doi: 10.1213/01.ane.0000250223.49963.0f. PMID 17179269
- [Background] Abdallah FW, Chan VW, Brull R. Transversus abdominis plane block: a systematic review. Reg Anesth Pain Med. 2012 Mar-Apr;37(2):193-209. doi: 10.1097/AAP.0b013e3182429531. PMID 22286518
- [Background] Yoshida T, Furutani K, Watanabe Y, Ohashi N, Baba H. Analgesic efficacy of bilateral continuous transversus abdominis plane blocks using an oblique subcostal approach in patients undergoing laparotomy for gynaecological cancer: a prospective, randomized, triple-blind, placebo-controlled study. Br J Anaesth. 2016 Dec;117(6):812-820. doi: 10.1093/bja/aew339. PMID 27956680
- [Background] Dai C, Zhang K, Huang J. The Efficacy of Transversus Abdominis Plane Block for Abdominal Hysterectomy Post-operative Analgesia. Cureus. 2018 Aug 10;10(8):e3131. doi: 10.7759/cureus.3131. PMID 30345190
- [Background] Easterday CL, Grimes DA, Riggs JA. Hysterectomy in the United States. Obstet Gynecol. 1983 Aug;62(2):203-12. PMID 6408544
- [Background] American Society of Anesthesiologists Task Force on Acute Pain Management. Practice guidelines for acute pain management in the perioperative setting: an updated report by the American Society of Anesthesiologists Task Force on Acute Pain Management. Anesthesiology. 2012 Feb;116(2):248-73. doi: 10.1097/ALN.0b013e31823c1030. No abstract available. PMID 22227789
- [Background] Chou R, Gordon DB, de Leon-Casasola OA, Rosenberg JM, Bickler S, Brennan T, Carter T, Cassidy CL, Chittenden EH, Degenhardt E, Griffith S, Manworren R, McCarberg B, Montgomery R, Murphy J, Perkal MF, Suresh S, Sluka K, Strassels S, Thirlby R, Viscusi E, Walco GA, Warner L, Weisman SJ, Wu CL. Management of Postoperative Pain: A Clinical Practice Guideline From the American Pain Society, the American Society of Regional Anesthesia and Pain Medicine, and the American Society of Anesthesiologists' Committee on Regional Anesthesia, Executive Committee, and Administrative Council. J Pain. 2016 Feb;17(2):131-57. doi: 10.1016/j.jpain.2015.12.008. PMID 26827847